CLINICAL TRIAL: NCT05105373
Title: Implementation Science and Impact Evaluation of PfR Programme: A Hybrid cRCT Design
Acronym: UPRISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Glasgow (Other); Oak Foundation (Other); Network of European Foundations (Unknown); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Uprise2021
Record Dates: First submitted 2021-09-30; First posted 2021-11-03 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Parenting; Gender-based Violence; Child Maltreatment; IPV

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial Hybrid Type 2 Evaluation
Who Masked: Participant, Outcomes Assessor
Masking Description: The allocation status of other participating families will be concealed from participants, thus reducing the potential for contamination. Research assistants conducting data assessments and statisticians conducting analysis will be blind to allocation in order to minimise assessment bias. Different groups of research assistants will be employed for outcome assessments and monitoring of implementation fidelity and adherence. Any instances of compromised blinding will be immediately reported. In the case of instances of harm or severe abuse being reported by a participant at any stage of the study, the allocation status of the participant will be un-blinded. All cases of un-blinding will be reported. Because of facilitators' involvement in the programme implementation, blinding will not be possible for service providers. Similarly, of course, participants cannot be blind to their own treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Parenting for Respectability (Experimental): Randomisation in the cRCT will be conducted at the cluster level. PfR is a 16-session manualised programme starting with nine single sex sessions followed by seven mixed sex sessions, delivered once a week by two local facilitators who receive one week's training. Activities were developed specifically for PfR or adapted from other parenting programs, including Project H, Stepping Stones, Mema kwa Jamii, The International Child Development Programme and Parenting for Lifelong Health. The programme addresses four familial processes associated with GBV and VAC: poor parental bonding and child attachment; harsh parenting; inequitable socialisation by gender and parental conflict. A particular goal is to involve fathers, whom most parenting programmes find hard to recruit, and the first nine sessions are delivered in single-sex groups.
  Interventions: Behavioral: Parenting for Respectability
- Control-Parenting for Respectability in a nutshell (Active Comparator): Randomisation in the cRCT will be conducted at the cluster level immediately after baseline data collection. Parents allocated to the control arm will receive a two-hour structured lecture called Parenting in a Nutshell on parenting and partner relationships. Three topics will be covered: 1) child development; 2) positive parenting; and 3) resolving partner conflicts. Facilitators delivering this lecture will have same/similar expertise with the facilitators engaged in PfR. .
  Interventions: Behavioral: Parenting for Respectability

INTERVENTIONS:
Behavioral: Parenting for Respectability — The programme addresses main challenges of Parenting and builds skills in 4 main areas
  1. Poor parental bonding and child attachment;
  2. Harsh parenting
  3. Inequitable socialisation by gender
  4. Parental conflict.

SUMMARY:
The Implementation science and impact evaluation of PfR programme: A hybrid cRCT design study will use an effectiveness-implementation hybrid type 2 design to a) determine the effectiveness and cost-effectiveness of PfR, and b) determine the feasibility and impact of three different implementation strategies in terms of programme delivery. A cluster randomised controlled trial (cRCT) will examine the effectiveness, cost-effectiveness, and implementation of the Parenting for Respectability (PfR) programme on the reduction of violence against children and gender based violence in comparison to those receiving an hour lecture on parenting in the Wakiso and Amuru districts of Uganda (N = 54 clusters, 2,160 parents, 1,080 children, 1:1 allocation ratio).

DETAILED DESCRIPTION:
Intimate partner violence (IPV) and violence against children (VAC) are interlinked and are major social, development and public health concerns. Globally it is estimated that approximately 30% ever-partnered women worldwide have experienced physical and/or sexual violence by an intimate partner at some point in their lives. IPV prevalence among women in Uganda is very high. The Uganda Demographic and Health Survey 2018 found that 36% of women had ever experienced partner physical violence, while 22% had ever experienced partner sexual violence. Violence against children is extremely widespread globally, with approximately half of all children - one billion aged 2-17 years - reporting having experienced violence in the past year. Furthermore, one in five women and up to one in ten men have been victims of sexual violence in childhood. The Uganda national VAC survey 2015 found that 59% girls and 68% boys had experienced physical violence in their childhood, and 35% girls and 17% boys had experienced sexual violence in their childhood. Such violence in Uganda and most Sub-Saharan African countries is usually perpetrated by people known to children in their homes and community. IPV and VAC are major causes of morbidity and mortality, they undermine the social functioning of the victims and their families, and have lifetime consequences for physical, sexual, reproductive and mental health. The prevention of both forms of violence would contribute to many Sustainable Development Goals since they strain health systems, lower educational achievement and economic productivity, and undermine economic and social development, and elimination of IPV is essential to Goal Five.

Many studies confirm the link between VAC and IPV, suggesting the need for an integrated approach to their prevention. A recent narrative review identified six ways in which they are interrelated: they have many shared risk factors, starting in the family; social norms legitimise both and discourage children and women from seeking help; both often occur within the same household both can be transmitted across generations; they can have similar consequences across the lifespan, and finally, both intersect in adolescence, a time of heightened vulnerability to violence.

Factors perpetuating IPV and VAC exist at multiple socio-ecological levels. For IPV, familial level factors include having been abused as a child, having an absent or rejecting father, inter-partner conflict, and male control of wealth and decision-making. Community level factors include women's isolation and male peer groups that legitimize men's violence. At the macro level IPV is associated with cultural norms that condone violence within the family, schools and community, establish rigid gender roles and link masculinity to toughness, male honour, dominance and ownership of women, and it thrives where policy, legislation and implementation of laws is weak. VAC is more likely in families that have difficulties developing stable, warm and positive relationships, where parents are unresponsive to their children, have harsh or inconsistent parenting styles, believe that corporal punishment is an acceptable form of discipline or have a poor understanding of child development, and therefore unrealistic expectations about the child's behaviour.

Recognizing that IPV is perpetuated at multiple levels, preventative interventions often focus on other psychosocial problems, e.g. poverty or alcohol abuse, as well as on inter-partner violence, although they are more effective if their main aim is to reduce IPV. The shared familial risk factors for IPV and VAC, and the increasing policy interest in optimizing parenting influence, provides a great opportunity for early intervention. An increasing number of parenting programs are being implemented and tested in LMICs to reduce VAC, and evidence is emerging that, if delivered by trained lay workers, they can be effective in improving child outcomes. However, interventions directly addressing early prevention of both IPV and VAC in LMICS remain limited.

Furthermore, very few parenting programs in LMICs harness cultural drivers and pre-existing motivations to change behaviour. In sub-Saharan Africa little attention has been paid to one of the most important dimensions of parenthood for both mothers and fathers: the need to maintain the family's respectability, in large part achieved through the appropriate behaviour of the children and their parents. This core motivation might be harnessed in the design of interventions to reduce spousal violence, modify negative parenting and encourage sensitive parenting, in order to reduce children's future risk of sexual, physical and/or emotional violence. In Uganda, the investigators are not aware of any parenting programs that deliberately recruit parental couples to complete both single and mixed sex sessions. The Investigators therefore designed a community-based parenting program, - Parenting for Respectability (PfR), - to address this gap in Uganda, and contribute evidence on how a parenting program can address both IPV and VAC. Following careful formative evaluation, the investigators conducted a pre-post study to establish whether there was sufficient evidence of effectiveness to warrant progression to a randomized controlled trial.

The programme has undergone formative evaluation (2014-16), 'Proof of Concept' pre-post outcome evaluation (2016-2019), and with support from Evaluation Fund, is currently being evaluated to assess implementation and scale-up modalities (April 2020-October 2021) in central Uganda. The investment in developing PfR so far has provided important lessons about the acceptability of PfR and how to refine it. Preliminary outcome evidence suggests that a rigorous evaluation of PfR is warranted. The pre-post study has found significant change across primary outcomes for both parent- and child-reports, including large effects for reduced harsh parenting (Cohen's f2 = 0.42, p < .001) and dysfunctional spousal relationships (Cohen's f2 = 0.28, p < .001), as well as increased positive parenting (Cohen's f2 = 0.48, p < .001). The programme has been disseminated widely in Uganda (www.parenting.ug.org), and both government and NGOs have expressed interest to scale it. However, two key uncertainties remain: (i) the optimal way to scale up the intervention in a 'real-world setting', and (ii) whether the evidence of effectiveness would be confirmed through a more rigorous, experimental, evaluation. As a result, this study will combine a rigorous cluster randomised control trial (cRCT) evaluation of PfR with an implementation study using a hybrid type 2 design to examine its effectiveness and cost-effectiveness as well as answer critical contextually relevant implementation science questions. This is essential to ensure that precious resources are not wasted and that there are no harmful unintended consequences from the programme.

ELIGIBILITY:
Inclusion criteria for participating parents or caregivers:

1. Age 18 or older;
2. Primary caregiver responsible for the care of a child between the ages of 10 and 14;
3. Agreement to participate in the PfR programme if allocated to the treatment condition;
4. Provision of consent to participate in the full study.

Inclusion criteria for participating children:

1. Age 10 to 14 years;
2. Live in the same household as primary caregiver who is part of PfR study;
3. Parent/caregiver gives consent to participate in the study;
4. Provision of consent to participate in the full study.

Inclusion criteria for facilitators:

1. Age 18 or older;
2. Facilitator who is involved in the delivery of the Parenting for Respectability programme;
3. Provision of consent to participate in the full study.

inclusion criteria for community development officers

1. Age 18 or older;
2. Involvement in delivery of PfR, or existing leadership role in communities where PfR is delivered;
3. Provision of consent to participate in the full study.

Exclusion Criteria:

Exclusion criteria for participating parents or caregivers:

1. Below Age 18;
2. Not a Primary caregiver responsible for the care of a child between the ages of 10 and 14;
3. Does not Provide consent to participate in the full study.

Exclusion criteria for participating children:

1. Below Age 10 and above age 14
2. Does not Live in the same household as primary caregiver who is part of PfR study;
3. Parent/caregiver does not gives consent to participate in the study;

Exclusion criteria for facilitators:

1. Below age 18;
2. Facilitator who is Not involved in the delivery of the Parenting for Respectability programme;
3. Does not Provide consent to participate in the full study.

Exclusion criteria for community development officers

1. Below age 18;
2. Is not Involved in the delivery of PfR, or has no existing leadership role in communities where PfR is delivered;
3. Does not provide consent to participate in the full study

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3162 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Assessing a Change in Child maltreatment - physical and emotional abuse; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child maltreatment will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (17 items, ICAST-Trial).
Assessing a Change in Child maltreatment - physical and emotional abuse; Child Report on Male Parent Figure | Baseline, 8-months post-baseline and 12-months post-baseline
  Child maltreatment will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (13 items, ICAST-Trial).
Assessing a Change in Child maltreatment - physical and emotional abuse; Child Report on Female Parent Figure | Baseline, 8-months post-baseline and 12-months post-baseline
  Child maltreatment will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (13 items, ICAST-Trial).
Assessing a Change in Intimate partner violence - perpetration; Parent-report | Baseline, 8-months post-baseline and 12-months post-baseline
  Perpetration of intimate partner violence (parent-report) will be measured using adapted versions of the Revised Conflict Tactics Scale Short Form (6 items; CTS2S).
Assessing a Change in Intimate partner violence -victimisation; Parent-report | Baseline, 8-months post-baseline and 12-months post-baseline
  Intimate partner violence victimisation (parent-report) will be measured using adapted versions of the Revised Conflict Tactics Scale Short Form (6 items; CTS2S).
Assessing a Change in Partner conflict; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Partner conflict will be assesses using a Revised Conflict Tactics Short Form based on two items assessing dysfunctional adult relationships in the household (e.g., "Your parents/carers or any other adults in your household quarrelled or had verbal arguments with each other").

SECONDARY OUTCOMES:
Assessing a Change in Child physical abuse-Parent report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child physical abuse will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (7 items, ICAST-Trial).
Assessing a Change in Child physical abuse; Child Report on Male Parent Figure | Baseline, 8-months post-baseline and 12-months post-baseline
  Child physical will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (5 items, ICAST-Trial).
Assessing a Change in Child physical abuse; Child Report on Female Parent Figure | Baseline, 8-months post-baseline and 12-months post-baseline
  Child physical will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (5 items, ICAST-Trial).
Assessing a Change in Child emotional abuse; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child emotional abuse will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (10 items, ICAST-Trial)
Assessing a Change in Child emotional abuse; Child Report on Male Parent Figure | Baseline, 8-months post-baseline and 12-months post-baseline
  Child emotional abuse will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (8 items, ICAST-Trial).
Assessing a Change in Child emotional abuse; Child Report on Female Parent Figure | Baseline, 8-months post-baseline and 12-months post-baseline
  Child emotional abuse will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (8 items, ICAST-Trial).
Assessing a Change in Child neglect; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child neglect will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (2 items, ICAST-Trial).
Assessing a Change in Child neglect; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child neglect will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (4 items, ICAST-Trial).
Assessing a Change in Community physical and sexual violence; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Children's experience of physical and sexual violence in the community in the past month will be based on one item (e.g., "In the past month, how often did adults in your community such as teachers, employer religious or community leaders, neighbours and other adults kick, punch, beat or threaten you with a knife or any other weapon physically?". Responses will be based on a Likert scale ranging from 0=Never to 3=Often.
Assessing a Change in Child sexual abuse; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child sexual abuse will be measured using an adapted version of the ISPCAN Child Abuse Screening Tool-Trial scale (10 items, ICAST-Trial).
Assessing a Change in Intimate partner coercion- perpetration; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Intimate partner coercion perpetration (parent-report) will be measured using an adapted version of the WHO questionnaire on women's health and life events.
Assessing a Change in Intimate partner coercion - victimisation; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Intimate partner coercion victimisation (parent-report) will be measured using an adapted version of the WHO questionnaire on women's health and life events
Assessing a Change in Intimate partner psychological aggression - perpetration; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Psychological aggression (parent-report) will be measured an adapted version of the Revised Conflict Tactics Scale Short Form (2 items; CTS2S).
Assessing a Change in Intimate partner psychological aggression - victimisation; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Psychological aggression victimisation (parent-report) will be measured using an adapted version of the Revised Conflict Tactics Scale Short Form (2 items; CTS2S).
Assessing a Change in Intimate partner physical aggression - perpetration; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Physical aggression perpetration (parent-report) will be measured using an adapted version of the Revised Conflict Tactics Scale Short Form (4 items; CTS2S).
Assessing a Change in Intimate partner physical aggression - victimisation; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Physical aggression victimisation (parent-report) will be measured using an adapted version of the Revised Conflict Tactics Scale Short Form (4 items; CTS2S).
Assessing a Change in Intimate partner sexual violence - perpetration; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Physical aggression perpetration (parent-report) will be measured using an adapted version of the Revised Conflict Tactics Scale Short Form (2 items; CTS2S).
Assessing a Change in Intimate partner sexual violence - victimisation; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Intimate partner sexual violence victimisation (parent-report) will be measured an adapted version of the Revised Conflict Tactics Scale Short Form (2 items; CTS2S).
Assessing a Change in Attitudes toward punishment; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Attitudes toward punishment will be assessed using two items based on the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module.
Assessing a Change in Attitudes toward punishment; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Attitudes toward punishment will be assessed using one item from the UNICEF Multiple Indicator Cluster Survey (MICS) 5 Child Discipline module.
Assessing a Change in Partner negotiation; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Partner negotiation will be based on four items adapted from the Revised Conflict Tactics Scale Short Form (9 items; CTS2S).
Assessing a Change in Positive partner relationships; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Positive partner relationships witnessed by children will be based on one item (e.g., "In the past month, how often did your parent figures in your household say nice things to each other in your presence?").
Assessing a Change in Positive parenting; Adult Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Positive parenting will be assessed using 10 items adapted from the Alabama Parenting Questionnaire (APQ-SF).
Assessing a Change in Positive parenting; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Positive parenting will be assessed using 20 items adapted from the Alabama Parenting Questionnaire (APQ-SF).
Assessing a Change in Parental monitoring; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Parental monitoring will be assessed using 6 items adapted from the Alabama Parenting Questionnaire (APQ-SF)
Assessing a Change in Parental monitoring; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Parental monitoring will be assessed using 10 items adapted from the Alabama Parenting Questionnaire (APQ-SF).
Assessing a Change in Educational aspirations; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Educational aspirations will be measured by one item asking the parent, "How far would you like your child to go in school?" rated on a 5-point scale
Assessing a Change in Educational aspirations; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Educational aspirations will be measured by one item asking the child, "How far would you like to go in school?" rated on a 5-point scale
Assessing a Change in Educational expectations; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Educational expectations will be measured using one item asking the parent how far they think their child will actually go in school rated on the same 5-point scale.
Assessing a Change in Educational expectations; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Educational expectations will be measured using one item asking the child how far they think they will actually go in school rated on the same 5-point scale.
Assessing a Change in Educational re-enrolment; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Educational re-enrolment will be assessed for children who are not currently in school by asking parents whether or not they would want them to go back to school. (0=No, 1=Yes)
Educational re-enrolment; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Educational re-enrolment will be assessed for children who are not currently in school by asking children whether or not they would want to go back to school (0=No, 1=Yes).
Assessing a Change in Parent support of education; Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Parental support for school will be measured by asking how often the parent engages in behaviours that support learning using a 5-point Likert scale
Assessing a Change in Parent support of education; Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Parental support for school will be measured by asking how often the child's male and female parent figures engage in behaviours that support learning using a 5-point Likert scale.
Assessing a Change in Child behaviour problems; Adult Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child behaviour problems will be measured using the Child and Adolescent Behaviour Inventory (CABI). 0 = Not True; 1 = Somewhat or Sometimes true; 2 = Very True; 999=Refused to answer; 888=Not Applicable. 19 items
Assessing a Change in Child behaviour problems: Child and Adolescent Behaviour Inventory - Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child behaviour problems will be measured using the Child and Adolescent Behaviour Inventory (CABI). 0 = Not True; 1 = Somewhat or Sometimes true; 2 = Very True; 999=Refused to answer; 19 items.
Assessing a Change in Child substance use - Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child substance use will be measured using two items based on lifetime alcohol and tobacco consumption (e.g. "Have often do you drink alcohol?"). Responses will be based on a 4-point Likert scale of 0 to 3 (0=Never; 3=Often).
Assessing a Change in Child prosocial behaviour - Adult Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child prosocial behaviour will be assessed from items derived from the pre-post study of PfR (5 items; e.g."Your child is considerate of other people's feelings.").
Assessing a Change in Child prosocial behaviour - Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child prosocial behaviour will be assessed from items derived from the pre-post study of PfR (5 items; e.g., "You are considerate of other people's feelings.")
Assessing a Change in Child respectful behaviour - Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Respectful behaviour by children will be assessed by asking parents one question about how often they see their children behaving well.
Assessing a Change in Gender socialisation - Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Gender socialisation of children will be assessed based on asking parents whether they agree or disagree about a series of statements regarding gender roles.
Assessing a Change in Gender socialisation - Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Gender socialisation of children will be assessed based on asking children whether they agree or disagree about a series of statements regarding gender roles.
Assessing a Change in Respectability - Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Respectability will be assessed by asking parents two questions regarding their attitudes to parental responsibilities regarding respectability.
Assessing a Change in Respectability - Child Report | Baseline, 8-months post-baseline, and 12-months post-baseline
  Respectability will be assessed by asking children eight questions regarding parental behaviour enforcing and modelling respectability.
Assessing a Change in Parenting stress - Parent Report | Baseline, 8-months post-baseline, and 12-months post-baseline
  Parenting stress (parent-report) will be based on a reduced version of the Parenting Stress Scale (9 items; PSS).
Assessing a Change in Adult depression - Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Adult depression (parent-report) will be measured using the depression subscale from the Depression, Anxiety, and Stress Scale.e,g. "How often in the past week, have you felt sad or down?").
Assessing a Change in Adult experience of violence during childhood - Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Adult experience of violence during childhood will be assessed using 6 items covering a range of childhood exposure to violence.
Assessing a Change in Communication about Sexual Behaviour - Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Communication about sexual behaviour by parents will be assessed by asking caregivers whether or not they have engaged in conversations with their children about puberty and sexual reproductive health.
Assessing a Change in Communication about Sexual Behaviour - Child Report | Baseline, 8-months post-baseline and 12-months post-baseline
  Child report of communication about sexual behaviour by parents will be assessed by asking caregivers whether or not their male and female parent figures have engaged in conversations with them about puberty and sexual reproductive health.
Assessing a Change in Impact of COVID-19 - Parent Report | Baseline, 8-months post-baseline and 12-months post-baseline
  The impact of COVID-19 will be assessed by asking parents to indicate whether they have been stressed by Covid-19, whether the child has been affected by Covid-19 and where the spouse relationship has been affected by Covid-19 agree.

OTHER OUTCOMES:
Adult experience of violence during childhood - Parent Report | Baseline
  Adult experience of violence during childhood will be assessed using 6 items covering a range of childhood exposure to violence, including witnessing partner conflict to experiencing corporal punishment and sexual abuse.
Basic childhood necessities - Parent Report | Baseline
  Relative poverty will be assessed using an adapted version of the Basic Necessities Scale (6 items). Developed by the Centre for South African Social Policy in the 'Indicators of Poverty and Social Exclusion Project.
Basic childhood necessities - Child Report | Baseline
  Relative poverty will be assessed using an adapted version of the Basic Necessities Scale (6 items). Developed by the Centre for South African Social Policy in the 'Indicators of Poverty and Social Exclusion Project.
Family stressors - Parent Report | Baseline
  Family stressors will be based on six items measuring the presence or absence of the following challenging situations in each household.
Food insecurity - Adult Report | Baseline
  Food insecurity will be assessed by asking adult respondents to report on whether their household was able to provide meals at breakfast, lunch, and dinner in the past month based on a Likert scale (0 =No; 1=Yes, sometimes; 2=Yes, always).
Food insecurity - Child Report | Baseline
  Food insecurity will be assessed by asking child respondents to report on whether their household was able to provide meals at breakfast, lunch, and dinner in the past month based on a Likert scale (0 =No; 1=Yes, sometimes; 2=Yes, always).
Basic caregiver and child demographic information - Child and Adult Report | Baseline
  Basic caregiver and child demographic information will be asked using items from the UNICEF Multiple Indicators Cluster Survey (MICS) Household Survey.
Recruitment rate - Assessor Report | 8-months post-baseline
  Recruitment rate will be based on the number of families who were eligible for inclusion and provided consent to participate in the program divided by the number of target population who were exposed to recruitment activities.
Enrolment rate - Facilitator Report | 8-months post-baseline
  Enrolment rate will be based on the number of families who attend either at least one session of Parenting for Respectability or the Parenting in a Nutshell lecture divided by the number of families allocated to either study arm.
Participation rate - Parenting for Respectability participants only - Facilitator Report | 8-months post-baseline
  Participation rates for those allocated to the PfR programme will be mean attendance rate for programme sessions based on those families who enrolled in the programme.
Dropout rate - Facilitator Report | 8-months post-baseline
  Dropout rates for enrolled participants will be defined as the percentage of participants who fail to attend at least three consecutive sessions and do not attend any sessions at a later stage.
Completion rate - Facilitator Report | 8-months post-baseline
  Completion rates for participants will be determined based on the number of enrolled participants who attend a cut-off threshold of at least 62.5% of the programme (i.e., 10 sessions)
Implementation dosage (time) - Facilitator Report | 8-months post-baseline
  Facilitators will report on the start and end time of each session/lecture in their weekly reports. Implementation dosage will be based on the total amount of time delivered divided by the mean attendance rate.
Time cost for delivery - Facilitator Report | 8-months post-baseline
  Time cost for delivery will be collected from facilitator weekly reports and based on the time spent on training, preparation, travel to and from, and delivery of each session/lecture.
Implementation fidelity - Facilitator Report | 8-months post-baseline
  Implementation fidelity by programme facilitators of the PfR programme will be examined using self-report checklists by the programme facilitators.
Competent adherence - Observational | 8-months post-baseline
  Competent adherence will be assessed using the PfR Facilitator Assessment Tool (PfR-FAT).
Qualitative Outcomes - In-depth Interviews | 8-months post-baseline, 12-months post-baseline
  In-depth interviews with senior implementation staff (N=4)
Qualitative Outcomes - Focus Group Discussions | 8-months post-baseline, 12-months post-baseline
  The researchers will have Focus group discussions with caregivers (N=8, 10 per FGD).
Qualitative Outcomes - Semi Structured Interviews | 8-months post-baseline, 12-months post-baseline
  Data will be collected through semi-structured interviews with Wakiso and Amuru District Community Development Services (N=4)
Cost effectiveness data collection | 8-months post-baseline, 12-months post-baseline
  Programme costs will be calculated using a micro-costing approach.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Godfrey Siu, PHD, Principal Investigator — Child Health and Development Centre, Makerere University; Dr. Jamie M. Lachman, D.PHIL, Principal Investigator — University of Glasgow: MRC/CSO Social and Public Health Sciences Unit
Locations (1):
- Wakiso Busukuma and Amuru Lamogi subcounties, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT05105373/Prot_000.pdf